CLINICAL TRIAL: NCT04230057
Title: Pharmacokinetics Study of Antitumor B in Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Ming Hu, Professor, University of Houston
Other Study IDs: STUDY00001235
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Healthy Adults
Keywords: Pharmacokinetics; Antitumor B; healthy volunteer
MeSH Terms: interventions — Antitumor B; antitumor A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteer: * In good general health and feeling well (no diagnosed disorders/illnesses)
  * At least 18 years old
  * BMI in the range of 18-29.9 kg/m²
  * No known history of substance abuse
  * No known allergies to food/drug
  Interventions: Dietary Supplement: Antitumor B

INTERVENTIONS:
Dietary Supplement: Antitumor B — Single dose 2400 mg
  Other Names: Zeng Sheng Ping; ACAPHA; ATB

SUMMARY:
The purpose of this study is to evaluate the single-dose oral pharmacokinetics of an herbal supplement - Antitumor B - in healthy subjects.

DETAILED DESCRIPTION:
Antitumor B (ATB), also known as Zeng Sheng Ping, is a Chinese herbal mixture composed of six plants: Sophora tonkinensis, Polygonum bistorta, Prunella vulgaris, Sonchus brachyotus, Dictamnus dasycarpus, and Dioscorea bulbifera. ATB is available as 300 mg tablets and has been traditionally used in China for dysplasia (dose 4-8 tables/ twice daily). Several studies in rodents and humans have been published demonstrating the chemopreventive activity of ATB against various cancers (e.g. lung, esophageal and oral). However, the investigators currently do not know what pharmacologically relevant concentration levels can be achieved systemically for different components of ATB in humans. Since it is a complex herbal mixture containing various key active components (KACs), relative levels of KACs in the ATB mixture can influence the bioavailability and pharmacokinetic of the individual KACs. The proposed study aim to estimate the plasma concentration of four key active components in a tablet with a chemical-defined ATB mixture. The investigators are interested in doing a human single-dose (8 tablets once) full pharmacokinetic study of ATB tablets. The investigators plan to collect 9 blood and 9 saliva samples from 8 healthy volunteers over a period of 24 hours (at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours) to

1. determine the saliva and plasma concentration of four key constituents of ATB (matrine, dictamnine, maackiain, fraxinellone) and
2. develop the in vivo correlation between plasma and saliva concentrations

ELIGIBILITY:
Inclusion Criteria:

* A potential subject must meet all the following inclusion criteria to be eligible to participate in the study.

  1. Health questionnaire filled on the day of recruitment, after signing the written consent form
  2. Participants must receive administration of study agent within 21-28 calendar days of being selected as subject after screening procedure is completed
  3. Healthy male or female subjects aged ≥18 and ≤40 years of age
  4. Subjects must have a body mass index (BMI) between 18.0-29.9 kg/m² inclusive
  5. CBC/differential obtained within 14 calendar days prior to selection as subject for drug administration , with adequate bone marrow function defined as follows: Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3; Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb

     ≥ 8.0 g/dl is acceptable.);
  6. Adequate renal and hepatic function within 14 calendar days prior to selection as subject for drug administration defined as follows: Serum creatinine < 1.5 mg/dl or creatinine clearance (CCr) ≥ 50 ml/min within 14 calendar days prior to selection as subject for drug administration, determined by 24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)
  7. Total bilirubin < 2 x the institutional Upper limit of Normal range (ULN) within 14 calendar days prior to selection as subject for drug administration
  8. AST or ALT ≤ 3 x the institutional ULN within 14 calendar days prior to selection as subject for drug administration
  9. ALP or GGT ≤ 2.5 x the institutional ULN within 14 calendar days prior to selection as subject for drug administration
  10. Magnesium, calcium, glucose, potassium, and sodium within 14 calendar days prior to selection as subject for drug administration, with the following required parameters: Magnesium: > 0.9 mg/dl or < 3 mg/dl; Calcium: > 7 mg/dl or < 12.5 mg/dl; Glucose: > 40 mg/dl or < 250 mg/dl; Potassium: > 3 mmol/L or < 6 mmol/L; Sodium: > 130 mmol/L or < 155 mmol/L.
  11. Participant must have active health insurance coverage at the time of study
  12. Participants must be able to understand study-specific information and instructions in English.
  13. Participant must be willing to fully comply with study procedures and restrictions.
  14. Participant must be able to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (1996) and applicable regulations, before completing any studyrelated procedures

Exclusion Criteria:

1. History of active liver disease or cancer.
2. Severe current or recurrent comorbidity such as (e.g., cardiovascular, haematological, neurological, endocrine, renal, liver, GI, HIV-AIDS, or other conditions such as cancer) that could affect the absorption and/or disposition of ATB
3. Any disease/illness diagnosed by a licensed physician.
4. Blood report positive for HIV and/or Hepatitis B and C tests
5. Has had an acute illness within two weeks prior to screening.
6. Pregnant or lactating women are ineligible due to unforeseeable risks to embryo or fetus.
7. Concurrent use of any prescription medication (including medicinal botanical) except birth control pills, over the counter medication and supplements except Vitamins and mineral supplements, or herbal supplements in form of herbal mixtures, teas or individual compounds (such as querctein, curcumin, echinacea, flaxseed, ginseng, ginkgo, soy etc.) that the study PI believes could potentially impact the results/objectives of this study.
8. Concurrent use of recreational drugs or alcohol during the study (self-declared by study participants)
9. Prisoners
10. Economically and/or educationally disadvantaged persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects in University of Houston and nearby area
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Cmax of matrine, dictamnine, maackiain and fraxinellone in plasma | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose
  Maximum (peak) observed drug concentration in plasma
Cmax of matrine, dictamnine, maackiain and fraxinellone in saliva | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose
  Maximum (peak) observed drug concentration in saiva
Tmax of matrine, dictamnine, maackiain and fraxinellone in plasma | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose
  Time of Maximum (peak) observed drug concentration in plasma
Tmax of matrine, dictamnine, maackiain and fraxinellone in saliva | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose
  Time of Maximum (peak) observed drug concentration in saliva
AUC0-24 of matrine, dictamnine, maackiain and fraxinellone in plasma | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose
  Area under the curve of plasma concentration-time profile
AUC0-24 of matrine, dictamnine, maackiain and fraxinellone in saliva | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose
  Area under the curve of saliva concentration-time profile

SECONDARY OUTCOMES:
Plasma-saliva IVIVC | Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours post dose
  In vivo-in vivo correlation established between plasma and saliva concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hu, PhD, Principal Investigator — University of Houston
Locations (1):
- University of Houston, College of Pharmacy, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin PZ, Zhang JS, Cao SG, Rong ZP, Gao RQ, Han R, Shu SP. [Secondary prevention of esophageal cancer--intervention on precancerous lesions of the esophagus]. Zhonghua Zhong Liu Za Zhi. 1988 May;10(3):161-6. Chinese. PMID 3219974
- [Background] Lin P, Zhang J, Rong Z, Han R, Xu S, Gao R, Ding Z, Wang J, Feng H, Cao S. Studies on medicamentous inhibitory therapy for esophageal precancerous lesions--3- and 5-year inhibitory effects of antitumor-B, retinamide and riboflavin. Proc Chin Acad Med Sci Peking Union Med Coll. 1990;5(3):121-9. PMID 2098764
- [Background] Lin P. [Medicamentous inhibitory therapy of precancerous lesions of the esophagus--3 and 5 year inhibitory effect of antitumor B, retinamide and riboflavin]. Zhongguo Yi Xue Ke Xue Yuan Xue Bao. 1990 Aug;12(4):235-45. Chinese. PMID 2147582
- [Background] Sun Z, Guan X, Li N, Liu X, Chen X. Chemoprevention of oral cancer in animal models, and effect on leukoplakias in human patients with ZengShengPing, a mixture of medicinal herbs. Oral Oncol. 2010 Feb;46(2):105-10. doi: 10.1016/j.oraloncology.2009.06.004. Epub 2009 Dec 21. PMID 20022553
- [Background] Zhang Z, Wang Y, Yao R, Li J, Yan Y, La Regina M, Lemon WL, Grubbs CJ, Lubet RA, You M. Cancer chemopreventive activity of a mixture of Chinese herbs (antitumor B) in mouse lung tumor models. Oncogene. 2004 May 6;23(21):3841-50. doi: 10.1038/sj.onc.1207496. PMID 15021904
- [Background] Wang Y, Yao R, Gao S, Wen W, Du Y, Szabo E, Hu M, Lubet RA, You M. Chemopreventive effect of a mixture of Chinese Herbs (antitumor B) on chemically induced oral carcinogenesis. Mol Carcinog. 2013 Jan;52(1):49-56. doi: 10.1002/mc.20877. Epub 2011 Nov 15. PMID 22086836
- [Background] Yin T, Yang G, Ma Y, Xu B, Hu M, You M, Gao S. Developing an activity and absorption-based quality control platform for Chinese traditional medicine: Application to Zeng-Sheng-Ping(Antitumor B). J Ethnopharmacol. 2015 Aug 22;172:195-201. doi: 10.1016/j.jep.2015.06.019. Epub 2015 Jun 20. PMID 26099633
- [Background] Gao S, Yang Z, Yin T, You M, Hu M. Validated LC-MS/MS method for the determination of maackiain and its sulfate and glucuronide in blood: application to pharmacokinetic and disposition studies. J Pharm Biomed Anal. 2011 May 15;55(2):288-93. doi: 10.1016/j.jpba.2011.01.015. Epub 2011 Jan 22. PMID 21349678
- [Background] Yang Z, Gao S, Yin T, Kulkarni KH, Teng Y, You M, Hu M. Biopharmaceutical and pharmacokinetic characterization of matrine as determined by a sensitive and robust UPLC-MS/MS method. J Pharm Biomed Anal. 2010 Apr 6;51(5):1120-7. doi: 10.1016/j.jpba.2009.11.020. Epub 2009 Nov 26. PMID 20034755
- See also: Standardization and Clinical Testing of ACAPHA for Cancer Prevention Part 1 of 3 — https://www.youtube.com/watch?v=IByBdYGRQig
- See also: Standardization and Clinical Testing of ACAPHA for Cancer Prevention Part 2 of 3 — https://www.youtube.com/watch?v=qmRewC7kkcU
- See also: Standardization and Clinical Testing of ACAPHA for Cancer Prevention Part 3 of 3 — https://www.youtube.com/watch?v=jMXDUFo5LoE
- See also: ACAPHA in Preventing Lung Cancer in Former Smokers With Bronchial Intraepithelial Neoplasia — https://clinicaltrials.gov/ct2/show/NCT00522197?term=acapha&rank=1